CLINICAL TRIAL: NCT02329353
Title: Clinical And Microbiological Analysis Of Orally Administered Lactobacillus Probiotic Lozenges In Chronic Periodontitis Patients Among Smokers And Non-smokers And Its Correlation With Clinical Parameters - A Clinico-Microbiological Study
Brief Title: Effect of Probiotics on Chronic Periodontitis in Smoker and Non- Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Next Gen Pharma India Pvt. Ltd. (Industry)
Collaborators: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAN_PERIO-SOM_01
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoker group (Experimental): 30 chronic periodontitis patients, having habit of smoking, with probing pocket depth of equal or greater than 5 mm with bleeding on probing and radio-graphic evidence of bone loss in at at least 2 sites at each quadrant will be given three probiotic lozenge per day for 8 weeks
  Interventions: Drug: Lactobacillus brevis CD2 Lozenges
- Non-smoker (Experimental): 30 chronic periodontitis patients, not having habit of smoking, with probing pocket depth of equal or greater than 5 mm with bleeding on probing and radio-graphic evidence of bone loss in at at least 2 sites at each quadrant will be given three probiotic lozenge per day for 8 weeks
  Interventions: Drug: Lactobacillus brevis CD2 Lozenges

INTERVENTIONS:
Drug: Lactobacillus brevis CD2 Lozenges — Each lozenge contains not less than 1 billion Colony forming unit of Lactobacillus brevis CD2
  Other Names: Probiotics

SUMMARY:
Periodontitis is one of the most common chronic inflammatory disease with the etiology of bacterial plaque and is associated with a number of putative bacterial species. The periodontal destruction is substantially mediated by the host, driven by the bacterial challenge. The presence of pathogenic bacteria with the absence of so-called "beneficial bacteria" and the susceptibility of the host are the main aetiological factors of periodontal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients free from any systemic illness
* Previously untreated moderate to severe generalised chronic periodontitis.
* Patients free from adverse reactions to lactose or fermented milk products
* Patient unwilling to quit smoking and smokers over the past one year ( Smoker arm).

Exclusion Criteria:

* Previous history of antibiotic usage over past 6 months
* Patients who are eligible for antibiotic usage during the treatment course
* Patients who are pregnant, lactating, alcoholic or who had undergone any surgical or nonsurgical therapy within 6 months.
* Acute oral lesions or necrotising ulcerative periodontitis

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Clinical Periodontal Indices | 8 weeks
  Improvement in clinical periodontal indices, namely, Plaque Index (PI), Gingival Index (GI), Probing Pocket Depth (PPD)

SECONDARY OUTCOMES:
Change in microbiological indices | 8 weeks
  Porphyromonas gingivalis, Tanerella forsythus

CONTACTS AND LOCATIONS:
Overall Officials: Rudrakshi chickanna, MDS, Principal Investigator — KRISHNADEVARAYA COLLEGE OF DENTAL SCIENCES AND HOSPITAL, BANGALORE; Shruthi J R, BDS, Principal Investigator — KRISHNADEVARAYA COLLEGE OF DENTAL SCIENCES AND HOSPITAL, BANGALORE; Prabhuji MLV, MDS, Principal Investigator — KRISHNADEVARAYA COLLEGE OF DENTAL SCIENCES AND HOSPITAL, BANGALORE
Locations (1):
- Krishnadevaraya College of Dental Sciences and Hospital, Bangalore, Karnataka, India